CLINICAL TRIAL: NCT03156738
Title: A Randomised, Double-blind, Placebo-controlled, Study to Investigate the Safety, Tolerability and Pharmacokinetics of Single Ascending Doses of MT-2990 in Healthy Male Subjects
Brief Title: A Clinical Study to Investigate How Safe and Tolerable the Study Drug MT-2990 is and How MT-2990 is Taken up by the Body in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: MT-2990-E01
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Dose 1 (Experimental): MT-2990 or Placebo
  Interventions: Drug: MT-2990; Drug: Placebo
- Dose 2 (Experimental): MT-2990 or Placebo
  Interventions: Drug: MT-2990; Drug: Placebo
- Dose 3 (Experimental): MT-2990 or Placebo
  Interventions: Drug: MT-2990; Drug: Placebo
- Dose 4 (Experimental): MT-2990 or Placebo
  Interventions: Drug: MT-2990; Drug: Placebo
- Dose 5 (Experimental): MT-2990 or Placebo
  Interventions: Drug: MT-2990; Drug: Placebo

INTERVENTIONS:
Drug: MT-2990 — Subjects will receive a single IV dose of MT-2990
Drug: Placebo — Subjects will receive a single IV dose of placebo

SUMMARY:
The purpose of this study is to investigate the safety, tolerability, pharmacokinetics and immunogenicity of MT-2990 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are able and willing to provide written informed consent to participate in this study
* Healthy male subjects aged 18 to 55 years (inclusive)
* Free from clinically significant (CS) illness or disease
* Body weight of 60 to 100 kg (inclusive)
* Body mass index (Quetelet index) ranging from 18 to 30 kg/m2 (inclusive).

Exclusion Criteria:

* A CS endocrine, thyroid, hepatic, respiratory, gastrointestinal, neurological (including history of seizures), renal, cardiovascular disease, or history of any significant psychiatric/psychotic illness or disorder (including anxiety, depression and reactive depression)
* Presence or history of any known malignancy with the exception of basal cell carcinoma in situ of the skin that has been treated with no evidence of recurrence within 6 months prior to the Screening Visit
* A history of bacterial or viral infections that led to hospitalisation and IV antibiotic or antiviral treatment within 3 months prior to Screening, or any recent infection requiring antibiotic or antiviral treatment within 4 weeks of Day -1
* A history of recurrent or chronic sinusitis, bronchitis, pneumonia, urinary tract infection (recurrent or chronic infection is two episodes within 6 months)
* A history of tuberculosis (TB) or malaria; history or any evidence of active infection or febrile illness within 7 days of dosing (e.g., bronchopulmonary, urinary, or gastrointestinal)
* An active, or history of, parasitic infections; any history of known or suspected congenital or acquired immunodeficiency state or condition that would compromise the subject's immune status (e.g., history of splenectomy)
* Presence or history of severe adverse reaction or allergy to any drug or allergy that is of clinical significance to the Investigational Medicinal Product (IMP)
* A positive test result for QuantiFERON-TB Gold® Plus, hepatitis B surface antigen, hepatitis B core antibody, hepatitis C antibody, or human immunodeficiency virus (HIV)-1 or HIV-2 antibodies at Screening.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2017-12-29 (Actual); Study Completion 2017-12-29 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as measured by incidence, nature and severity of adverse events | Up to Day 85
  Adverse events will be summarised by dose level.
Safety and tolerability as measured by vital signs | Up to Day 85
  Vital signs variables and changes from Baseline will be summarised by dose level.
Safety and tolerability as measured by ECG parameters | Up to Day 85
  12-lead ECG variables and changes from Baseline will be summarised by dose level.
Safety and tolerability as measured by clinical laboratory assessments | Up to Day 85
  Laboratory variables and changes from Baseline will be summarised by dose level.
Safety and tolerability as measured by physical examination | Up to Day 85
  Physical examination data will be listed by subject.

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) of MT-2990 | Up to Day 85
  Cmax will be summarised by dose level.
Measured time of maximum observed serum concentration (tmax) of MT-2990 | Up to Day 85
  tmax will be summarised by dose level.
Apparent terminal elimination half-life (t1/2) of MT-2990 | Up to Day 85
  t½ will be summarised by dose level.
AUC from time zero to the last measurable concentration (AUC0-last) of MT-2990 | Up to Day 85
  AUC0-last will be summarised by dose level.
AUC from time zero to infinity (AUC0-∞) of MT-2990 | Up to Day 85
  AUC0-∞ will be summarised by dose level.
Terminal elimination rate constant (Kel) of MT-2990 | Up to Day 85
  Kel will be summarised by dose level.
Apparent volume of distribution at steady state (Vss) of MT-2990 | Up to Day 85
  Vss will be summarised by dose level.
Apparent volume of distribution during terminal phase after IV administration (Vz) of MT-2990 | Up to Day 85
  Vz will be summarised by dose level.
Mean residence time from time zero to infinity (MRT0-∞) of MT-2990 | Up to Day 85
  MRT0-∞ will be summarised by dose level.
Apparent serum clearance (CL) of MT-2990 | Up to Day 85
  CL will be summarised by dose level.
Percentage of AUC obtained by extrapolation (%AUCex) of MT-2990 | Up to Day 85
  %AUCex will be summarised by dose level.
Proportion of subjects who develop antibodies against MT-2990 in serum | Up to Day 85
  The proportion of subjects who develop antibodies against MT 2990 in serum will be summarised using descriptive statistics on the Safety Analysis Set.

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (1):
- Pharmaceutical Research Associates (PRA) Health Sciences, NZ Groningen, Netherlands